CLINICAL TRIAL: NCT02613832
Title: Immediate Effect of Expiratory Positive Airway Pressure and Breath Stacking in Non-cooperative Patients Detected by Electrical Impedance Tomography
Brief Title: Applicability of Techniques of Lung Expansion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Caio César Araújo Morais, Specialist in cardiopulmonary physiotherapy, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Caio01
Record Dates: First submitted 2013-10-25; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Stroke
Keywords: Noncooperative patients
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPAP Group (Experimental): The EPAP devices increase the alveolar pressure. This effect is obtained through valves that generate a resistance to airflow during expiration.
  Interventions: Other: EPAP
- Breath Stacking Group (Experimental): The Breath Stacking consists on the implementation of subsequent inspiratory efforts through a one way valve, which allows stacked volume of gas during each inspiration, until it reaches a maximum lung volume.
  Interventions: Other: Breath Stacking

INTERVENTIONS:
Other: EPAP — The EPAP will be applied with a Spring Load Valve Resistor (Vital Signs, Totowa, NJ, USA), adjusted with a pressure of 10 cmH2O. The Spring Load Valve Resistor will be connected to the expiratory branch of the T-tube. Duration of intervention: 5 minutes.
  Other Names: Expiratory Positive Airway Pressure
  Arms: EPAP Group
Other: Breath Stacking — The BS will be performed by a T-tube with a one-way inspiratory valve and the expiratory branch occluded. The expiratory occlusion is maintain until observed the presence of a plateau in the impedance plethysmogram by EIT, which corresponds to the absence of inspired air displacement or when a maximum time of 40 seconds was attained. Durantion of intervention:Three BS interventions will be performed at one minute intervals between them.
  Other Names: Air Stacking
  Arms: Breath Stacking Group

SUMMARY:
The survival of patients with lesions in the central nervous system is usually accompanied by physical and mental sequelae. These impairments favor the prolonged restriction to the bed, which may contribute with changes in respiratory function. In this context, lung re-expansion techniques are used to prevent or treat the various respiratory complications.

DETAILED DESCRIPTION:
The survival of patients with lesions in the Central Nervous System is usually accompanied by physical and mental permanents sequelae. This impairment of cognitive status associated with motor injury favors prolonged restriction of these patients to the bed, which may contribute to the emergence of other health damages. In the clinical practice, lung expansion techniques has been used as a prophylaxis and treatment of respiratory conditions that involve volumetric reductions. However, the deficit of awareness and cooperation difficult the use of several therapeutic resources. There are few interventions that could be proposed due to no need the collaboration to be performed, such as Breath Stacking technique (BS) and Expiratory Positive Airway Pressure (EPAP). The BS is characterized by execution of inspiratory cycles through a one way valve, which allows stacked volume of gas during each inspiration, until it reaches values approximate to maximum inspiratory capacity. While in the EPAP, alveolar pressure is elevated to breath against a expiratory flow resistance generated by a spring load valve. The effects on lung volume promoted BS and EPAP can be safely measured using an electrical impedance tomography (EIT). This recent imaging modality offers information about lung air volumes distribution and have a strong linear correlation with regional ventilation within the thorax. The effects on lung volume promoted BS and EPAP can be safely measured using an EIT monitor. This recent imaging modality offers information about lung air volumes distribution and have a strong linear correlation with regional ventilation within the thorax. Until this moment, there is not description about the effect of lung expansion techniques on regional lung parameters.

ELIGIBILITY:
Inclusion criteria:

1. Patients undergoing neurosurgery restricted to bed for more than 14 days;
2. Aged between 18 and 65 years;
3. Glasgow Coma Scale < 10 points;
4. Breathing spontaneously through the tracheostomy tube;
5. No respiratory infection;
6. Chest circumference between 88 and 98 centimeters;

Exclusion criteria:

1. Presence of chronic lung diseases;
2. Chest deformity;
3. Rib fracture;
4. Asymmetrical chest expansion;
5. Abdomen distension;
6. Spasticity in any hemisphere with Ashworth Scale score more than 2 points for upper limbs;
7. Uncoordinated movements of the limbs;
8. Cardiorespiratory instability (heart rate < 60 or > 120 bpm; respiratory rate > 35 ipm; mean arterial pressure < 60 mmHg or > 120 mmHg; oxygen saturation < 90%).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Regional Lung Aeration | Before and 1, 5, 10, 15, 30, 60, 90, 120 minutes post-intervention.
  Change in Regional Lung Aeration (difference between the End-Expiratory Lung Impedance before and post-intervention). Each image along the time represent the relative change in impedance distribution within the transverse section of the chest, from the first scan (before intervention) to current scan. The pixel values are express as percentage changes of local impedance.

SECONDARY OUTCOMES:
Regional Lung Ventilation | Before and 1, 5, 10, 15, 30, 60, 90, 120 minutes post-intervention.
  Change in Regional Lung Ventilation (difference between end-inspiratory and end-expiratory lung impedance before and post-intervention).
Heart Rate | Before and 1, 5, 10, 15, 30, 60, 90, 120 minutes post-intervention.
  Change in Heart Rate (beats per minute).
Mean Arterial Pressure | Before and 1, 5, 10, 15, 30, 60, 90, 120 minutes post-intervention.
  Change in Mean Arterial Pressure (mmHg)
Respiratory Rate | Before and 1, 5, 10, 15, 30, 60, 90, 120 minutes post-intervention.
  Change in Respiratory Rate (breath per minute)
Periferic Saturation of Oxygen | Before and 1, 5, 10, 15, 30, 60, 90, 120 minutes post-intervention.
  Change in Periferic Saturation of Oxygen (fraction of oxygen-saturated hemoglobin relative to total hemoglobin).

CONTACTS AND LOCATIONS:
Overall Officials: Caio César A Morais, Master, Study Chair — Universidade Federal de Pernambuco; Shirley L Campos, PHD, Study Chair — Universidade Federal de Pernambuco
Locations (1):
- Hospital of Clinics of the Federal University of Pernambuco, Recife, PE - Pernambuco, Brazil

REFERENCES:
- [Background] Bayford R, Tizzard A. Bioimpedance imaging: an overview of potential clinical applications. Analyst. 2012 Oct 21;137(20):4635-43. doi: 10.1039/c2an35874c. PMID 22930423
- [Background] Costa EL, Lima RG, Amato MB. Electrical impedance tomography. Curr Opin Crit Care. 2009 Feb;15(1):18-24. doi: 10.1097/mcc.0b013e3283220e8c. PMID 19186406
- [Background] Victorino JA, Borges JB, Okamoto VN, Matos GF, Tucci MR, Caramez MP, Tanaka H, Sipmann FS, Santos DC, Barbas CS, Carvalho CR, Amato MB. Imbalances in regional lung ventilation: a validation study on electrical impedance tomography. Am J Respir Crit Care Med. 2004 Apr 1;169(7):791-800. doi: 10.1164/rccm.200301-133OC. Epub 2003 Dec 23. PMID 14693669
- [Background] Baker WL, Lamb VJ, Marini JJ. Breath-stacking increases the depth and duration of chest expansion by incentive spirometry. Am Rev Respir Dis. 1990 Feb;141(2):343-6. doi: 10.1164/ajrccm/141.2.343. PMID 2301851
- [Derived] Morais CC, Campos SL, Lima CS, Monte LJ, Bandeira MCP, Brandao DC, Costa EL, Aliverti A, Amato MB, Andrade AD. Acute Effects of Lung Expansion Maneuvers in Comatose Subjects With Prolonged Bed Rest. Respir Care. 2021 Feb;66(2):240-247. doi: 10.4187/respcare.07535. Epub 2020 Oct 6. PMID 33024002